CLINICAL TRIAL: NCT00670371
Title: Factors of Importance for the Subjective and Objective Burden of Informal Caregivers to Patients With Functional Psychoses - a Descriptive and Comparative Study
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Birgit Ekholm, MD, Medical Director Neuroscience, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-NSE-DUM-2007/1
Record Dates: First submitted 2008-04-29; First posted 2008-05-01 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Functional Psychoses; Informal Caregivers
Keywords: Caregiver burden
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Patients having the following diagnoses are eligible for inclusion into the study: schizophrenia, schizophreniform disorder, schizoaffective disorder, brief psychotic disorder, delusional disorder, affective psychosis with mood incongruent delusions, psychotic disorder not otherwise specified or patients being actively psychotic.
- 2: Closest relative(s) /informal caregiver(s)

SUMMARY:
The objective is to find determinants for the subjective and objective burden of informal caregivers to patients who are requiring continued antipsychotic treatment for functional psychoses among factors related to the patient, the health care and support provision system and the informal caregiver him/her-self.

DETAILED DESCRIPTION:
The study also comprises a descriptive part with the aim:

* To describe clinical characteristics, symptoms, and functioning in the patient group.
* To describe patient resource use in terms of support from the health care and social care sector.
* To describe the socio-economic situation, the general and psychological health, and the coping ability of the informal caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Patients, male or female, aged 18 years or more, suffering or having suffered from a psychotic episode and being in need of continuous antipsychotic medication.
* The respective patient must have at least one informal caregiver.
* Subjects (patients and informal caregivers) must be able to read and write.

Exclusion Criteria:

* Diagnosis of dementia and such cognitive impairment which makes self assessments even with assistance unreliable (patients and informal caregivers).
* Involvement in the planning and conduct of the study (patients and informal caregivers).
* Other concurrent medical condition interfering with ability to complete study (patients and informal caregivers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Psychiatric patients and informal caregivers. Selected from outpatient wards
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-03; Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Dencker Vansvik, Study Director — AstraZeneca, MC, Sweden; Lena Flyckt, Principal Investigator — Danderyds Hospital, Stockholm
Locations (9):
- Sweden (9):
  - Research site, Bromma
  - Research Site, Danderyd
  - Research Site, Falköping
  - Research Site, Huddinge
  - Research Site, Lidingö
  - Research Site, Ljungby
  - Research Site, Malmo
  - Research Site, Solna
  - Research Site, Stockholm